CLINICAL TRIAL: NCT04438759
Title: Clinical Efficacy of Virtual Reality for Acute Pain and Anxiety Management During Outpatient Hysteroscopy and Endometrial Biopsy in Subfertility Patients
Brief Title: Clinical Efficacy of Virtual Reality During Office Hysteroscopy and Endometrial Biopsy in Subfertility
Acronym: HYSVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYSVIR
Record Dates: First submitted 2020-02-28; First posted 2020-06-19 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: Infertility, Female
Keywords: virtual reality; hysteroscopy; infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: This study is a comparison between the current standard practice of performing a diagnostic hysteroscopy and a relatively recently developed technology that is added to the standard diagnostic hysteroscopy. The aim of the study is to find out whether this newer technology has an advantage for the patient, in the form of anxiety and pain reduction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational group (Experimental): Virtual Reality
  Interventions: Device: Oncomfort, commercially available Virtual Reality headset
- reference group (No Intervention): standard of care

INTERVENTIONS:
Device: Oncomfort, commercially available Virtual Reality headset — Virtual Reality headset, consisting of headphones with smartphone glasses - see oncomfort.com/en, CE approval conform 93/42/EEC and 2007/47/EEC
  Arms: investigational group

SUMMARY:
This study is a comparison between the current standard practice of performing a diagnostic hysteroscopy and a relatively recently developed technology that is added to the standard diagnostic hysteroscopy. The aim of the study is to find out whether this newer technology has an advantage for the patient, in the form of anxiety and pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* undergoing fertility treatments
* for which outpatient hysteroscopy has been prescribed
* for different possible indications: suspicion of intracavitary pathology, recurrent implantation failure, recurrent early pregnancy loss, …

Exclusion Criteria:

1. Hearing impairments and blindness
2. Motion sickness
3. Any known anatomical characteristics that may make performing the office procedure impossible.
4. The unwillingness of the patient to undergo an office hysteroscopy
5. Denial or withdrawal of informed consent

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — hysteroscopy requires presence of uterus
Enrollment: 216 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain experience as assessed using visual analog scale | 1/ baseline pre-procedure 2/ immediately after the procedure (1+2= day of office hysteroscopy) and 3/ 1 week after the procedure
  quantified through visual analog scale: from 0.0 to 10.0cm, ranging from 0.0 meaning 'No pain' and 10.0 representing 'worst imaginable pain'.

CONTACTS AND LOCATIONS:
Overall Officials: valerie schutyser, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel CRG, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No